CLINICAL TRIAL: NCT00959595
Title: Improvement of Sensibility in the Sole of the Foot in Diabetic Patients, Induced by EMLA-application to the Lower Leg - a Double Blind Study
Brief Title: Improvement of Sensibility in the Foot in Diabetic Patients Induced by EMLA-application to the Lower Leg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Goran Lundborg, Professor Göran Lundborg, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-001834-29
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; neuropathy; foot; sensibility; brain plasticity
MeSH Terms: conditions — Diabetes Mellitus | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMLA cream (Experimental)
  Interventions: Drug: EMLA cream
- Placebo cream (Placebo Comparator): A placebo cream identical in appearance and consistency to the experimental cream
  Interventions: Drug: EMLA cream

INTERVENTIONS:
Drug: EMLA cream — The study subjects are treated either by 50 g of a local anesthetic agent containing 2.5% Lidocaine and 2.5% Prilocaine (EMLA®, AstraZeneca - Södertälje, Sweden) or a placebo cream, applied to the lower leg. The cream is applied under occlusive bandage (plastic foam and a tube) for 1.5 hours circumferential to the lower leg 10-12 cm distally of the tibial tuberosity and the malleolus at ankle level. Administration of the treatment cream as well as removal after 1,5 hour and at sensory assessment after 1.5 hour and 24 hours, and interviewing the patient about subjective experience from the treatment are performed by an independent research nurse, not involved in the sensory assessment.
  Arms: EMLA cream
Drug: EMLA cream — 50g applied according to description of intervention

SUMMARY:
Sensory input from the foot as well as all other body parts results in activation of sensory cortex.

It is well known that the cortical body map is experienced-dependant and can rapidly change in response to changes in activity and sensory input from the periphery [10-12]. Increased activity and sensory input from the hand results in expansion of the cortical hand representation [13-15], while decreased sensory input, for instance by anaesthesia, amputation or nerve injury, results in shrinkage of the cortical hand representation [16-21]. Due to the constant ongoing "cortical competition" between body parts the adjacent cortical areas expand and take over the silent area, deprived of sensory input.

The investigators have recently described striking examples of such rapid cortical re-organisations induced by selective cutaneous anaesthesia of the forearm: application of EMLA cream to the volar aspect of the forearm results in improved sensory functions of the hand [18] linked to expansion of the hand representational area in sensory cortex . In analogy, EMLA application to the lower leg in healthy controls results in improved sensory functions in the sole of the foot linked to expansion of the foot representational area in sensory cortex.

To test the hypothesis that EMLA application to the lower leg of diabetic patients will result in improved sensory functions in the sole of the foot as well as expansion of the foot representation in sensory cortex. The investigators hypothesize that repeated applications of EMLA will result in a long lasting sensibility improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years) suffering from diabetes with subjective sensory impairment in the sole of the foot.

Exclusion Criteria:

* Patients with painful neuropathy or established ulcer formation in toes or sole of the foot, known hypersensitivity to local anaesthetics, major vascular reconstructions, communication problems due to severe language problems.
* Patients with pacemakers or magnetic implants or suffering from claustrophobia will not be subjected to fMRI-investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Touch thresholds in the sole of the foot (Semmes-Weinstein monofilaments) | Screening, before application, 90 min after application, 24 hours after application

SECONDARY OUTCOMES:
MRI | MRI-examination, before application, 90 min after application, 24 hours after application
fMRI | fMRI-examination, before application, 90 min after application, 24 hours after application

CONTACTS AND LOCATIONS:
Overall Officials: Göran Lundborg, Professor, Principal Investigator — Dpt of Hand Surgery, Malmö University Hospital, Lund University, Sweden
Locations (1):
- Department of Hand Surgery, Malmö University Hospital, Malmo, Sweden

REFERENCES:
- [Result] Lundborg GN, Bjorkman AC, Rosen BN, Nilsson JA, Dahlin LB. Cutaneous anaesthesia of the lower leg can improve sensibility in the diabetic foot. A double-blind, randomized clinical trial. Diabet Med. 2010 Jul;27(7):823-9. doi: 10.1111/j.1464-5491.2010.03014.x. PMID 20636964